CLINICAL TRIAL: NCT06242535
Title: Pilot Study of GLY-LOW Supplementation in Postmenopausal Women With Obesity
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hoskinson Health and Wellness Clinic (Industry)
Collaborators: Buck Institute for Research on Aging (Other); University of Wyoming (Other)
Responsible Party: Principal Investigator, Sanjay Dhar, Director of Research, Hoskinson Health and Wellness Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRANY IRB # 23-02-452-1498
Record Dates: First submitted 2024-01-29; First posted 2024-02-05 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Insulin Resistance; Obesity; Cardiovascular Diseases; Cognitive Impairment; Physical Disability; Depression; Inflammation; Hormone Deficiency; Physical Inactivity; Hyperlipidemias; Hypertension; Overeating
Keywords: nutrition supplement
MeSH Terms: conditions — Insulin Resistance; Obesity; Cardiovascular Diseases; Cognitive Dysfunction; Depression; Inflammation; Sedentary Behavior; Hyperlipidemias; Hypertension; Hyperphagia

STUDY DESIGN:
Intervention Model Description: One group, no-placebo comparer, pre post intervention clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- GLY-LOW supplement (Experimental): Each participant will take this supplement daily in a pill form orally once in the morning. The test product will be two capsules a day with breakfast between 7:00 - 11:00 AM. The chosen doses were based on dose conversion from mice to humans and the prior data on safety for each of the compounds in humans.
  Interventions: Biological: GLY-LOW

INTERVENTIONS:
Biological: GLY-LOW — This supplement is available for over-the-counter purchase. Each capsule is a combination of vitamins and natural products: Vitamin B1 (100mg); Vitamin B6 (50mg); Niacin (200mg); Alpha Lipoic Acid (150mg); and Piperine (15mg). The supplement, GLY-LOW, is FDA approved for use as a dietary supplement (IND 162006)
  Other Names: GLYLO

SUMMARY:
A combination of generally regarded as safe (GRAS) compounds named GLY-LOW, which included: alpha lipoic acid, pyridoxamine, nicotinamide, piperine and thiamine, were examined in pre-clinical experiments. GLY-LOW supplementation reduced caloric intake and increased insulin sensitivity in mice. In female mice, GLY-LOW supplementation reversed aging-related declines in female hormones. Studies in humans are needed to examine the feasibility, utility and efficacy of GLY-LOW supplementation in post-menopausal women with obesity toward improving aging-related impairments. The effect of GLY-LOW supplementation on these obesity and biological age-related impairments in post-menopausal adult female humans with obesity is unknown. We aim to translate the findings of GLY-LOW supplementation in animals to a cohort of healthy, postmenopausal females at birth with obesity by conducting a one-group, no-placebo comparer, pre post intervention clinical trial. Additionally, we propose to examine the specific effect of supplementation by GLY-LOW on biological aging via retina scan. The objectives of the proposed pilot study are:

I. Conduct a 6-month pilot study to examine the feasibility, utility and efficacy of GLY-LOW supplementation in a total of 40 postmenopausal female born adults > 55 years with obesity (≥ 30 BMI).

DETAILED DESCRIPTION:
Study Population:

Healthy, postmenopausal (> 1 year from last menstrual cycle) adult females (at birth), > 55 years of age with obesity (≥ 30 BMI)

Objectives/Purpose of the Study:

Worldwide rates of obesity increased from 100 million to 764 million between 1980 and 2021. During the same time frame, a five-fold increase in Type 2 diabetes (T2DM) was reported. Increases were similar across the globe with older individuals at greatest risk of obesity and related metabolic dysfunction. Central obesity is well known to be both a manifestation and driver of metabolic syndrome with similar prevalence worldwide. Older, post-menopausal females, in particular, are at increased risk of developing central obesity due to a reduction in endogenous ovarian hormone production. Novel multi-modal therapies are needed to address central obesity-related metabolic dysfunction in post-menopausal females. However, current therapeutic methods lack specificity and propose universal solutions to a multi-factorial disorder requiring an individualized, precision medicine approach. More concerning, is the lack of rigorous, scientific evidence to support conventional dietary therapies for reducing aging-related central obesity and associated metabolic dysfunction. Targeting multiple biological pathways that are related to individual behavioral determinants (caloric intake) and biological aging markers (estrogen levels) may identify more precise therapies in post-menopausal female adults with obesity.

Recently, advanced glycation end-products (AGEs) were identified as potential drivers of obesity-related impaired metabolic function. In a series of in vitro and in vivo experiments, a combination of GRAS compounds that function synergistically to improve metabolic health and extend lifespan [(alpha lipoic acid, pyridoxamine, nicotinamide, piperine and thiamine (i.e. GLY-LOW)] were examined. Supplementation with GLY-LOW was shown to detoxify methylglyoxal (MGO), a reactive precursor to AGEs. In addition, GLY-LOW supplementation reduced caloric intake and glycolysis, reprogramed metabolism, and increased insulin sensitivity and mTor signaling in the hypothalamus of the mice. In female animals GLY-LOW supplementation reversed aging-related declines in estrogen and related female hormones. Studies in humans are needed to translate these findings and explore the feasibility, utility and efficacy of GLY-LOW supplementation in post-menopausal women with obesity toward improving aging-related impairments. These include increased metabolic disease risk and insufficiency, impaired physical function, osteoporosis, reduced fitness levels, cognitive impairment, systemic inflammation and premature biological aging. Interestingly, results of a novel biological aging assessment, retina scan, were recently shown to be associated with metabolic dysfunction via inflammatory pathways. The effect of GLY-LOW supplementation on these obesity and biological age-related impairments in post-menopausal adult female humans with obesity is unknown.

Study Site:

The Hoskinson Health and Wellness Clinic (HHWC) focuses on your whole health for your whole life, and provides a proactive, not reactive, personalized and integrated, multi-component solution to age-related increases in obesity and associated declines in metabolic health. The HHWC utilizes functional, precision medicine to identify unhealthy aging biomarkers and genetic vulnerabilities, and innovative medical technology to both diagnose and manage aging-related metabolic, physical and cognitive impairments. State-of-the-art assessments identify targets for tailored programming including diet instruction, nutrition education and supplementation, fitness counseling and training. The HHWC proposes to conduct a series of clinical studies using these state-of-the-art measures of aging-related parameters. Initially, we aim to translate the findings of GLY-LOW supplementation in animals to a cohort of healthy, postmenopausal females at birth with obesity by conducting a one-group, no-placebo comparer, pre post intervention clinical trial. Additionally, we propose to examine the specific effect of supplementation by GLY-LOW on biological aging via retina scan. The objectives of the proposed pilot study are:

I. Conduct a 6-month pilot study to examine the feasibility, utility and efficacy of GLY-LOW supplementation in a total of 40 postmenopausal female born adults > 55 years with obesity (≥ 30 BMI)

Ia. Examine alterations in self-reported caloric intake and the following health and biological aging, parameters prior to and after 6 months of GLY-LOW supplementation:

1. Self-reported Caloric Intake
2. Metabolic disease risk
3. Cardiovascular disease risk
4. Metabolic assessments
5. Hormones
6. Physical Function and Fitness
7. Muscular strength
8. Cognitive Function and Depression assessments
9. Systemic inflammation
10. Biological aging
11. Safety parameters (also every 2 months during the intervention; ECG at baseline and 2 months only)
12. Compliance measures (pill counts and interviews every 2 months during the intervention)

Trial Design:

One group, no-placebo comparer, pre post intervention clinical trial

Randomization and Blinding:

The one group, no-placebo comparer pilot study will not require randomization. Study data managers and biostatisticians will be blinded to basic demographic and clinical characteristics (e.g. female, postmenopausal) of the study population and the overall purpose of the trial.

Initial Recruitment/Screening, Enrollment, and Baseline Evaluation:

Recruitment, screening and enrollment will occur during the first eight weeks of the study. Approximately 40 participants will be screened and enrolled into the study. Participation in the baseline evaluation will occur during weeks 9-12. Recruitment will be by referrals, personal interview, brochure mail-outs to area physicians, community center flyers and presentations, presentations at civic meetings, mass media announcements, social media posts, as well as clinic screenings as currently used in our existing studies and clinical services at the Hoskinson Health and Wellness Center. The plan is described below:

1. Potential study participants will be provided with a general information handout or link to our website regarding the study and contact information for participation.
2. Study personnel will receive phone, email inquiries or website inquiries and conduct a pre-screening interview and complete a checklist to determine eligibility.
3. Study personnel and/or other medical staff will then conduct the IRB-approved informed consent procedures and begin the screening process for study participants. An explanation of all procedures, potential risks, temporary side effects, anticipated benefits, and alternative methods (nutrition and fitness counseling, weight loss pharmaceuticals or nutraceuticals, other anti-aging therapeutics) will be given to the study participant. Confidentiality is assured as well as the right not to participate or to withdraw at any time. The signature of the study participant will be obtained on the consent form. A copy of the forms will be given to each study participant. Assurance that all questions have been answered about the study testing is obtained from the participants. Names and telephone numbers of contact persons on the medical team are given to each study participant for use if future questions arise.
4. General health screenings will then be performed by qualified medical staff. A medical physical evaluation to verify eligibility will be performed at the intervention baseline visits and a list of current medications will be required.
5. After clearance by the study physician, the study participant will receive the first set of baseline measurements The study coordinator will schedule the second day of baseline measurements with the study participant. The study participant will be advised to fast for at least 12 hours prior to the second day of baseline testing

Treatment, Dosage and Dosing regimen of the GLY-LOW supplement:

This supplement is available for over-the-counter purchase. Each capsule is a combination of vitamins and natural products: Vitamin B1 (100mg); Vitamin B6 (50mg); Niacin (200mg); Alpha Lipoic Acid (150mg); and Piperine (15mg). Each participant will take this supplement daily in a pill form orally once in the morning. The test product will be two capsules a day with breakfast between 7:00 - 11:00 AM. The chosen doses were based on dose conversion from mice to humans and the prior data on safety for each of the compounds in humans.

Expected Duration of Subject Participation:

34 weeks

Available Alternative Treatments:

Available alternative treatments offered at the HHWC include nutrition and fitness counseling, weight loss pharmaceuticals or nutraceuticals, other anti-aging therapeutics. Study participants will be provided with information concerning these alternative treatment therapies during the consent procedures.

Follow-up Assessments:

1. The study participant will attend a follow-up safety assessment visit every two months and will participate in blood tests and MSQ. ECG will be assessed at baseline and 2 months only.
2. The study participants will attend one follow-up assessment after 6 months of receiving the study supplement (GLY-LOW). Baseline measurements will be repeated during these follow-up assessments in order to examine the effectiveness of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal (>1 year from last menstrual cycle) adult females (at birth) >55 years of age with obesity (BMI ≥ 30)

Exclusion Criteria:

* Males
* Adults not females at birth
* Adult females diagnosed with Gout
* Adult females receiving hormone replacement therapy (HRT)
* Adult females who are currently prescribed or received weight loss medications within the past 6 months, or currently enrolled in a defined weight loss program.
* Adult females with cardio-metabolic disease [e.g. cardiovascular disease (CVD), type 2 diabetes (T2DM), hypertension, h/o stroke etc.)] requiring any prescription medication.
* Adult females with other chronic immune, pulmonary, neurodegenerative or systemic disease requiring prescription medication
* Adult females with severe asthma based upon American Thoracic Society (ATS) standards and/or NIH guidelines.
* Adult females requiring monoclonal antibody or biological treatment
* Adult females diagnosed with an acute lower respiratory or GI infection within 2 weeks
* Adult females who are pregnant (would not qualify as post-menopausal) or nursing mothers
* Adult females reporting moderate to severe mental or physical disability
* Adult females reporting unwillingness to travel to onsite clinical facilities
* Adult females with moderate to severe cognitive impairment
* Adult females diagnosed with an eating disorder
* Adult females on blood thinners and anti-platelet drugs (other than aspirin), on chronic steroids (including inhaled), on spironolactone, on statins, on diuretics, on chronic pain medications, on any medication that affects glucose, insulin, lipids, metabolic performance
* Adult females with any recent change in chronic disease or any recent change in medication.
* Adult females on supplements with potential to augment or compete with the GLY-LOW.

Min Age: 56 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Post-menopausal (>1 year from last menstrual cycle) adult females (at birth), >55 years of age with obesity (BMI ≥ 30)
Enrollment: 13 (Actual)
Dates: Start 2023-07-27 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Insulin Resistance (IR) | During the screening/baseline visit and again during the 6-month follow-up visit.
  Measured by examining biochemical markers using samples of whole blood obtained in a certified laboratory. . Study participants will be required to fast for 12 hours prior to the blood test. Blood collection and processing: Venous blood will be collected in the morning after a 12 hour fast with the study participant seated. Blood will be collected in tubes containing 1.5 mg/ml EDTA for procedures requiring plasma, in tubes with no additives for serum measures and citrate tubes for homeostasis endpoints.
Fasting Insulin (I) and Glucose (G) | During the screening/baseline visit and again during the 6-month follow-up visit.
  Measured by examining biochemical markers using samples of whole blood obtained in a certified laboratory. . Study participants will be required to fast for 12 hours prior to the blood test. Blood collection and processing: Venous blood will be collected in the morning after a 12 hour fast with the study participant seated. Blood will be collected in tubes containing 1.5 mg/ml EDTA for procedures requiring plasma, in tubes with no additives for serum measures and citrate tubes for homeostasis endpoints.
Glycosylated Hemoglobin [Hemoglobin A1C (HBA1C)] | During the screening/baseline visit and again during the 6-month follow-up visit.
  Measured by examining biochemical markers using samples of whole blood obtained in a certified laboratory. . Study participants will be required to fast for 12 hours prior to the blood test. Blood collection and processing: Venous blood will be collected in the morning after a 12 hour fast with the study participant seated. Blood will be collected in tubes containing 1.5 mg/ml EDTA for procedures requiring plasma, in tubes with no additives for serum measures and citrate tubes for homeostasis endpoints.
BMI [weight (kg) divided by height (m2)] | During the screening/baseline visit and again during the 6-month follow-up visit.
  Total body weight and height were measured with an electronically calibrated scale and stadiometer (Pelstart Health-o-meter Professional 500KL) with participants in light, loose fitting clothing without shoes.
Body Composition [lean mass, fat mass, bone density and area, central adiposity (DEXA); waist circumference] | During the screening/baseline visit and again during the 6-month follow-up visit.
  DEXA will be used for analysis of body composition using Hologics Horizon A DEXA. This machine is an FDA cleared-to market device. The procedure will be performed by trained technicians at the Hoskinson Health and Wellness Clinic. The study participants will be instructed to remove all metal and jewelry including their shoes before they are correctly positioned on the scan table, lying down on their back with their arms to their side. The DEXA will measure X-rays as they are transmitted through the study participant's body. The study participant will be exposed to ionizing radiation, but there is no discomfort during the measurement (0.02-0.03mR). This exposure is less than the 125mR/yr, which is the amount individuals receive from non-medical background radiation (Lunar). The low dose of radiation will not adversely affect the bone or surrounding tissue.

SECONDARY OUTCOMES:
Self-reported Caloric Intake | During the screening/baseline visit and again during the 6-month follow-up visit.
  Assessed using the ASA24-2022 Dietary Assessment Tool. Study participants will complete a 24hr food recall. Study personnel will download, process, and analyze the ASA24 data per NCI protocols.
Total Cholesterol, Low Density Lipoprotein (LDL), High Density Lipoprotein (HDL) and Triglycerides (TRI) | During the screening/baseline visit and again during the 6-month follow-up visit.
  Measured by examining biochemical markers using samples of whole blood obtained in a certified laboratory. . Study participants will be required to fast for 12 hours prior to the blood test. Blood collection and processing: Venous blood will be collected in the morning after a 12 hour fast with the study participant seated. Blood will be collected in tubes containing 1.5 mg/ml EDTA for procedures requiring plasma, in tubes with no additives for serum measures and citrate tubes for homeostasis endpoints. A small portion (approximately ½ teaspoon = 2.5 ml) of blood from the baseline and 6-month follow-up samples will be saved for future biomedical and molecular analysis.
Systolic (SBP) and Diastolic Blood Pressure (DPB) | During the screening/baseline visit and again during the 6-month follow-up visit.
  Resting SBP and DBP measured by a Welch Allen automated system. Two readings will be taken and averaged. If the two values differ by more than 5 mm Hg, an additional reading will be obtained. The study participant will abstain from eating and from heavy exercise for at least 2 hours prior to the test. Study participants will also be instructed not to ingest caffeine within 30 minutes before blood pressure measurements. The study participant will be comfortably seated, with the arm slightly flexed, palm up and the entire forearm supported at heart level on a smooth surface. Each measure will be directly recorded on the data spreadsheet in the study computer and the average score will be calculated by standard Microsoft functions.
Metabolic Assessments at Rest | During the screening/baseline visit and again during the 6-month follow-up visit.
  Resting energy expenditure (REE) and Respiratory Quotient (RQ) (Day 2) will be measured at rest.Individuals are instructed to fast for 12 hours prior to the test and are instructed not to engage in vigorous physical activity for 24 hours prior to the test. Individuals will be allowed to drink water prior to the test and will rest in a recumbent position for 30 minutes prior to the start of each testing session. Metabolic measurements will be continuously taken during the test. Expired gases will be sampled and analyzed for Volume of Oxygen (VO2) and Volume of Carbon Dioxide (VCO2) concentrations by indirect calorimetry calculated via a metabolic cart (Cosmed Quark CPET, Rome, Italy) using a canopy hood set up (Cosmed Quark RMR, Rome Italy).
Thyroid Stimulating Hormone (TSH), Follicle Stimulating Hormone (FSH), Luteinizing Hormone (LH), Estrogen (E) and Progesterone (P4) | During the screening/baseline visit and again during the 6-month follow-up visit.
  Measured by examining biochemical markers using samples of whole blood obtained in a certified laboratory. Study participants will be required to fast for 12 hours prior to the blood test. Blood collection and processing: Venous blood will be collected in the morning after a 12 hour fast with the study participant seated. Blood will be collected in tubes containing 1.5 mg/ml EDTA for procedures requiring plasma, in tubes with no additives for serum measures and citrate tubes for homeostasis endpoints. A small portion (approximately ½ teaspoon = 2.5 ml) of blood from the baseline and 6-month follow-up samples will be saved for future biomedical and molecular analysis.
Physical Function | During the screening/baseline visit and again during the 6-month follow-up visit.
  Measured by the short physical performance battery as follows:
  The short physical performance battery is comprised of three performance measures: 1) The standing balance test requires study participants to maintain their feet in a side-by-side, semi-tandem stand, or tandem stand for 10 seconds. 2) A test of walking speed where study participants walk for 4 minutes at a normal pace; 3) The chair stand test, which evaluates lower extremity extensor muscle strength by measuring the time required for the participants to stand up and sit down from a chair five times with arms folded across the chest. Each performance measure is scored from 1-4 points (maximum 12 points). This test can be accomplished in 15 minutes.
Muscular Strength | During the screening/baseline visit and again during the 6-month follow-up visit.
  Measured by administering the hand grip test as follows:
  The hand-grip strength procedure of the Hand-Held Dynamometer (Baseline) will be administered to patient participants seated in a chair with a back support and fixed arm rests using a calibrated instrument. The study participants will position their thumb around one side of the instrument and their fingers along the other side of the handle. They will be instructed to squeeze the handle as long and as tightly as possible. Three measures will be recorded for each hand, alternating sides. This procedure is shown to be a valid and feasible method of assessing muscular strength in elderly adults20-21.
Cardiorespiratory Fitness | During the screening/baseline visit and again during the 6-month follow-up visit.
  Measured by a graded submaximal treadmill test using a modified Balke protocol 22. A warm-up session of approximately 5 minutes will establish comfortable walking speeds. Study participants will then walk on the treadmill for 2-minute warm-up at 0% grade, the grade of the treadmill will then be increased by 2.5% every 2 minutes until the participant can no longer continue or reaches 80% of age-predicted volume of oxygen (VO2) peak. Following the warm-up session, VO2 and carbon dioxide VCO2 production, ventilation (VE) and respiratory exchange ratio (RER) will be calculated via a metabolic cart (Cosmed Quark CPET, Rome, Italy) and a two-way non-re-breathing mask (Cosmed K2 Mask, Rome, Italy).
Cognitive Function by the Mini-Mental State Examination (MMSE) | During the screening/baseline visit and again during the 6-month follow-up visit.
  The Mini Mental State Examination (MMSE) will be administered per standard protocol with the cut-off of 26. The MMSE is comprised of 30 questions that assesses cognitive function by evaluating attention and orientation, memory, registration, recall, calculation, language and ability to draw a complex polygon. The MMSE exhibits high levels of acceptance as a diagnostic instrument in both health care providers and researchers25. The MMSE is available in numerous language translations and can be administered in less than one hour.
Executive Function (EF), Cognitive Flexibility (CF) and Mental Control (MC) | During the screening/baseline visit and again during the 6-month follow-up visit.
  Measured by the Advanced Digital Cognitive Assessment of (BrainCheck28-29) which is a tablet-based version of six neurocognitive tests, which can be completed in 30 minutes: 1) Flanker Task, 2) Digit Symbol Substitution Test, 3) Stroop Task, 4) The Trail Making Test, 5) Balance and Coordination, 6) The Immediate and Delayed Recall Tests
Depression | During the screening/baseline visit and again during the 6-month follow-up visit.
  Measured by the Center for Epidemiologic Studies Depression Scale (CES-D Scale)30. Study participants are asked to read each question of a 20 item scale carefully, then circle one of the numbers to the right to indicate how they felt or behaved during the past week, including the assessment day. Options include: (0) Rarely or none of the time (less than 1 day), (1) Some or a little of the time (1-2 days), (2) Occasionally or a moderate amount of the time (3-4 days), (3) Most or all of the time (5-7 days). The test can be completed in approximately 10 minutes. The responses are totaled by the test administrator and the possible range of scores is between 0 to 60. Higher scores indicate the presence of more symptomatology of depression.
Systemic Inflammation | During the screening/baseline visit and again during the 6-month follow-up visit.
  assessed by measuring serum pro-and-anti- inflammatory markers, which will be obtained by simple blood draw as described above and evaluated by Enzyme Linked Immunoassay (ELISA); the panel will measure pro- and anti-inflammatory factors and cytokines previously shown to be associated with metabolic disease, obesity and aging. These include: C-Reactive Protein (hs-CRP). Blood samples will then be stored at -70 degrees Celsius in a freezer at the HHWC. The blood samples will then be shipped to the Buck Institute/USF for analysis. A commercially available kit for sTNFR1 human ELISA kit (Biosource international, CA) will be utilized.
Total Body Weight | During the screening/baseline visit and again during the 6-month follow-up visit.
  Measured with an electronically calibrated scale (Pelstart Health-o-meter Professional 500KL) will be used to obtain the weight in kilograms of each study participant. The study participant will remove her shoes and step on the scale. The study participant will remain as still as possible. The study participant's weight in kilograms will be recorded once the digital reading is constant. The study participant will remain on the scale until the weight is recorded. The process will be repeated two additional times.
Height | During the screening/baseline visit and again during the 6-month follow-up visit.
  Measured with a calibrated stadiometer (Pelstart Health-o-meter Professional 500KL) will be used to obtain the height in centimeters of each study participant. The study participant will remove her shoes and step onto the floor platform facing in an outward direction with the heels together. The scapula and buttocks will remain in contact with the back of the stadiometer during the measure. The head will be positioned in a horizontal plane. The clinician will move the headboard onto the most superior aspect of the study participant's head. This procedure will be repeated two additional times. The average height in to the nearest tenth of a centimeter (0.1 cm) will be calculated on the data statistical form.
Waist Circumference | During the screening/baseline visit and again during the 6-month follow-up visit.
  Measured in study participants with a tape measure. The measurement of girth at the waistline provides an estimation of central adiposity17. Individuals will wear light clothing for this measurement. They are asked to stand erect and in an upright position with abdomen relaxed, arms at sides and feet together. Measures are made at the end of normal expiration at the umbilicus. The measurements are recorded to the nearest 0.1 cm. This process is repeated and the average of each of the two circumferences is used in analysis (a third measurement is obtained if the first two measurements are greater than 0.5 cm apart). Figure 1 provides a graphic representation of the measurement site for waist circumference.
Biological Aging | During the screening/baseline visit and again during the 6-month follow-up visit.
  Biological Aging (Day 2) will be measured by retina scan to quantify biological aging (Welch Allyn® RetinaVue® 700 Imager) via standard clinical procedures.
Phenotypic Age | During the screening/baseline visit and again during the 6-month follow-up visit.
  Phenotypic age will be measured by blood test

OTHER OUTCOMES:
Safety Outcomes | During the screening/baseline visit, 2-, 4-, and 6-month follow-up visits.
  Safety outcomes include: 1) measurement of Thyroid Stimulation Hormone (TSH), Follicle-Stimulating Hormone (FSH), Luteinizing Hormone (LH) and blood platelet counts, 2) measurement of cardiac function by Electrocardiogram (ECG), 3) administration of the medical symptoms questionnaire (MSQ)
Subject adherence | During 2-, 4-, and 6-month follow-up visits.
  Trained clinical research staff interviewed participants about supplement intake, forgetfulness, and barriers to adherence. Staff reviewed supplement details, addressed side effects and concerns, and answered questions. Monitoring via pill counts were additional indicators of adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Dhar, PhD, Principal Investigator — Hoskinson Health and Wellness Clinic
Locations (1):
- Hoskinson Health and Wellness Clinic, Gillette, Wyoming, United States

IPD SHARING:
Plan to Share IPD: Yes
Data is available upon request.

REFERENCES:
- [Background] Hoskinson W, Sothern M, Thompson T, et al. 516 Follicle-stimulating hormone is reduced following a novel nutritional therapeutic in postmenopausal women with obesity. Journal of Clinical and Translational Science. 2025;9(s1):151-152. doi:10.1017/cts.2024.1097
- [Background] O'Hearn M, Lara-Castor L, Cudhea F, Miller V, Reedy J, Shi P, Zhang J, Wong JB, Economos CD, Micha R, Mozaffarian D; Global Dietary Database. Incident type 2 diabetes attributable to suboptimal diet in 184 countries. Nat Med. 2023 Apr;29(4):982-995. doi: 10.1038/s41591-023-02278-8. Epub 2023 Apr 17. PMID 37069363
- [Background] Jayedi A, Soltani S, Motlagh SZ, Emadi A, Shahinfar H, Moosavi H, Shab-Bidar S. Anthropometric and adiposity indicators and risk of type 2 diabetes: systematic review and dose-response meta-analysis of cohort studies. BMJ. 2022 Jan 18;376:e067516. doi: 10.1136/bmj-2021-067516. PMID 35042741
- [Background] Noubiap JJ, Nansseu JR, Lontchi-Yimagou E, Nkeck JR, Nyaga UF, Ngouo AT, Tounouga DN, Tianyi FL, Foka AJ, Ndoadoumgue AL, Bigna JJ. Geographic distribution of metabolic syndrome and its components in the general adult population: A meta-analysis of global data from 28 million individuals. Diabetes Res Clin Pract. 2022 Jun;188:109924. doi: 10.1016/j.diabres.2022.109924. Epub 2022 May 15. PMID 35584716
- [Background] Nappi RE, Chedraui P, Lambrinoudaki I, Simoncini T. Menopause: a cardiometabolic transition. Lancet Diabetes Endocrinol. 2022 Jun;10(6):442-456. doi: 10.1016/S2213-8587(22)00076-6. Epub 2022 May 4. PMID 35525259
- [Background] Brennan AM, Standley RA, Yi F, Carnero EA, Sparks LM, Goodpaster BH. Individual Response Variation in the Effects of Weight Loss and Exercise on Insulin Sensitivity and Cardiometabolic Risk in Older Adults. Front Endocrinol (Lausanne). 2020 Sep 10;11:632. doi: 10.3389/fendo.2020.00632. eCollection 2020. PMID 33013705
- [Background] Tamura Y, Omura T, Toyoshima K, Araki A. Nutrition Management in Older Adults with Diabetes: A Review on the Importance of Shifting Prevention Strategies from Metabolic Syndrome to Frailty. Nutrients. 2020 Nov 1;12(11):3367. doi: 10.3390/nu12113367. PMID 33139628
- [Background] Chaudhuri J, Bains Y, Guha S, Kahn A, Hall D, Bose N, Gugliucci A, Kapahi P. The Role of Advanced Glycation End Products in Aging and Metabolic Diseases: Bridging Association and Causality. Cell Metab. 2018 Sep 4;28(3):337-352. doi: 10.1016/j.cmet.2018.08.014. PMID 30184484
- [Background] Chaudhuri J, Bose N, Gong J, Hall D, Rifkind A, Bhaumik D, Peiris TH, Chamoli M, Le CH, Liu J, Lithgow GJ, Ramanathan A, Xu XZS, Kapahi P. A Caenorhabditis elegans Model Elucidates a Conserved Role for TRPA1-Nrf Signaling in Reactive alpha-Dicarbonyl Detoxification. Curr Biol. 2016 Nov 21;26(22):3014-3025. doi: 10.1016/j.cub.2016.09.024. Epub 2016 Oct 20. PMID 27773573
- [Background] Zee T, Bose N, Zee J, Beck JN, Yang S, Parihar J, Yang M, Damodar S, Hall D, O'Leary MN, Ramanathan A, Gerona RR, Killilea DW, Chi T, Tischfield J, Sahota A, Kahn A, Stoller ML, Kapahi P. alpha-Lipoic acid treatment prevents cystine urolithiasis in a mouse model of cystinuria. Nat Med. 2017 Mar;23(3):288-290. doi: 10.1038/nm.4280. Epub 2017 Feb 6. PMID 28165480
- [Background] Zhu Z, Liu D, Chen R, Hu W, Liao H, Kiburg K, Ha J, He S, Shang X, Huang Y, Wang W, Yu H, Yang X, He M. The Association of Retinal age gap with metabolic syndrome and inflammation. J Diabetes. 2023 Mar;15(3):237-245. doi: 10.1111/1753-0407.13364. Epub 2023 Mar 14. PMID 36919192